CLINICAL TRIAL: NCT03724500
Title: Clinical Significance of Circulating Tumor Cell in Non Small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CGMH-IRB-104-8753B
Record Dates: First submitted 2018-10-23; First posted 2018-10-30 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2023-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non small cell lung cancer; Circulating tumor cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
From literature review, circulating tumor cell was demonstrated its possible role in disease relapse. It was rare nit could be identified in all lung cancer patients. In addition, circulating tumor cell usual aggregate to form circulating tumor micro-emboli and caused distant metastases. Therefore, circulating tumor cell could play a role in detect disease relapse and appropriate treatment could be given more earlier and further prolong patients' survival. However, the detail clinical significance of circulating tumor still remain unknown. The aim of this study was evaluate the clinical significance, including present timing, numbers, and correlation to disease relapse, of circulating tumor cell in lung cancer patients. Investigators want to clarify the clinical significance between circulating tumor cell and clinical presentation of lung cancer in order to establish new prediction model and improve lung cancer patients' survival.

DETAILED DESCRIPTION:
Lung cancer was a major cause of cancer-related death worldwide. According to statistical data from Ministry of Health and Welfare, the incidence of lung cancer related death was 25.5 per 100,000 population. According to NCCN guideline, the standard treatment for patients with resectable disease is anatomic resection and mediastinal lymph node dissection. The current prognostic system, TNM system, was based of patho-histologic characteristics and this system provide the most important information about disease-free and overall survival for corresponding disease severity. According to investigators previous studies, investigators've identified risk factors for all lung cancer patients with resectable disease and poor prognostic factors in different TNM stage. Investigators could utilized factors that designed for all patients as an initial survey and further subgroup patients into high or low risk for relapse in subsequent stratification that utilized grading system in different TMN stage. If investigators could identified high risk patients, more aggressive treatment and follow up program may decreased risk of disease relapse and prolong patient survival.

From literature review, circulating tumor cell was demonstrated its possible role in disease relapse. It was rare nit could be identified in all lung cancer patients. In addition, circulating tumor cell usual aggregate to form circulating tumor micro-emboli and caused distant metastases. Therefore, circulating tumor cell could play a role in detect disease relapse and appropriate treatment could be given more earlier and further prolong patients' survival. However, the detail clinical significance of circulating tumor still remain unknown. The aim of this study was evaluate the clinical significance, including present timing, numbers, and correlation to disease relapse, of circulating tumor cell in lung cancer patients. Investigators want to clarify the clinical significance between circulating tumor cell and clinical presentation of lung cancer in order to establish new prediction model and improve lung cancer patients' survival.

ELIGIBILITY:
Inclusion Criteria:

1. Non-small cell lung cancer patients with stage I to III
2. Patients with resectable suspicious pulmonary malignant lesion

   1. no pre-operation diagnosis ( patients refused biopsy or difficult for biopsy)
   2. image survey showed clinical stage I to III

Exclusion Criteria:

1. Final pathology coexisted with small cell lung cancer component
2. Patients who presented as stage IIIb or IV.
3. Not received curative intended surgery due to multi-comorbidities.
4. Patients who presented in tumor seeding or positive resection in the final pathology
5. Patients who received neoadjuvant therapy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a resectable malignant or suspicious malignant pulmonary lesion
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Variation trend of circulating tumor cell counts | 1. Circulating tumor cell counts in pre-op, post-op, post-operation day 1 and post-operation day 3 ; 2.need complete 5-years surveillance (disease status confirmation)
  Relationship between variation trend of circulating tumor cells and disease relapse in patients with a suspicious pulmonary lesion after tumor resection

SECONDARY OUTCOMES:
Malignancy prediction capacity of circulating tumor cell counts | Pre-operation circulating tumor cells ( sampled before operation at operation day)
  Relationship between pre-operation circulating tumor cell counts and malignancy

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hsun Hsieh, MD, Principal Investigator — Chang Gung Memorial Hospital; Yi-Cheng Wu, MD, Principal Investigator — Chang Gung Memorial Hospital; Cheng-Ta Yang, MD, Principal Investigator — Chang Gung Memorial Hospital; JUI-YING Fu, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Background] Fernandes G, Sucena M, Lombardia E, Machado A, Hespanhol V, Queiroga H. Non small cell lung cancer - comparison between clinical and pathological staging. Rev Port Pneumol. 2006 Jul-Aug;12(4):337-57. English, Portuguese. PMID 16969567
- [Background] McCann J. PET scans approved for detecting metastatic non-small-cell lung cancer. J Natl Cancer Inst. 1998 Jan 21;90(2):94-6. doi: 10.1093/jnci/90.2.94. No abstract available. PMID 9450567
- [Background] Vaz AP, Fernandes G, Souto Moura C, Bastos P, Queiroga H, Hespanhol V. Integrated PET/CT in non small cell lung cancer staging--clinical and pathological agreement. Rev Port Pneumol. 2012 May-Jun;18(3):109-14. doi: 10.1016/j.rppneu.2012.01.004. Epub 2012 Mar 8. English, Portuguese. PMID 22405953
- [Background] Wu CY, Fu JY, Wu CF, Hsieh MJ, Liu YH, Wu YC, Yang CT, Tsai YH. Survival Prediction Model Using Clinico-Pathologic Characteristics for Nonsmall Cell Lung Cancer Patients After Curative Resection. Medicine (Baltimore). 2015 Nov;94(45):e2013. doi: 10.1097/MD.0000000000002013. PMID 26559298
- [Background] Wu CY, Fu JY, Wu CF, Liu YH, Hsieh MJ, Wu YC, Yang CT, Tsai YH. Pathologic Stage of Nonsmall Cell Lung Cancer Patients Presenting as Resectable Cases After Neoadjuvant Therapy Did Not Predict the Prognosis. Medicine (Baltimore). 2015 Oct;94(40):1. doi: 10.1097/MD.0000000000001700. PMID 26448022
- [Background] Wu CF, Fu JY, Yeh CJ, Liu YH, Hsieh MJ, Wu YC, Wu CY, Tsai YH, Chou WC. Recurrence Risk Factors Analysis for Stage I Non-small Cell Lung Cancer. Medicine (Baltimore). 2015 Aug;94(32):e1337. doi: 10.1097/MD.0000000000001337. PMID 26266381
- [Background] Wu CF, Wu CY, Fu JY, Wang CW, Liu YH, Hsieh MJ, Wu YC. Prognostic value of metastatic N1 lymph node ratio and angiolymphatic invasion in patients with pathologic stage IIA non-small cell lung cancer. Medicine (Baltimore). 2014 Oct;93(20):e102. doi: 10.1097/MD.0000000000000102. PMID 25365403
- [Background] Hsieh CP, Fu JY, Liu YH, Yang CT, Hsieh MJ, Tsai YH, Wu YC, Wu CY. Prognostic factors in resectable pathological N2 disease of non-small cell lung cancer. Biomed J. 2015 Jul-Aug;38(4):329-35. doi: 10.4103/2319-4170.145765. PMID 25432594
- [Background] Tognela A, Spring KJ, Becker T, Caixeiro NJ, Bray VJ, Yip PY, Chua W, Lim SH, de Souza P. Predictive and prognostic value of circulating tumor cell detection in lung cancer: a clinician's perspective. Crit Rev Oncol Hematol. 2015 Feb;93(2):90-102. doi: 10.1016/j.critrevonc.2014.10.001. Epub 2014 Oct 12. PMID 25459665
- [Background] Tanaka F, Yoneda K, Kondo N, Hashimoto M, Takuwa T, Matsumoto S, Okumura Y, Rahman S, Tsubota N, Tsujimura T, Kuribayashi K, Fukuoka K, Nakano T, Hasegawa S. Circulating tumor cell as a diagnostic marker in primary lung cancer. Clin Cancer Res. 2009 Nov 15;15(22):6980-6. doi: 10.1158/1078-0432.CCR-09-1095. Epub 2009 Nov 3. PMID 19887487
- [Background] Pantel K, Speicher MR. The biology of circulating tumor cells. Oncogene. 2016 Mar 10;35(10):1216-24. doi: 10.1038/onc.2015.192. Epub 2015 Jun 8. PMID 26050619
- [Background] Yoon SO, Kim YT, Jung KC, Jeon YK, Kim BH, Kim CW. TTF-1 mRNA-positive circulating tumor cells in the peripheral blood predict poor prognosis in surgically resected non-small cell lung cancer patients. Lung Cancer. 2011 Feb;71(2):209-16. doi: 10.1016/j.lungcan.2010.04.017. Epub 2010 May 14. PMID 20471712
- [Background] O'Flaherty JD, Gray S, Richard D, Fennell D, O'Leary JJ, Blackhall FH, O'Byrne KJ. Circulating tumour cells, their role in metastasis and their clinical utility in lung cancer. Lung Cancer. 2012 Apr;76(1):19-25. doi: 10.1016/j.lungcan.2011.10.018. Epub 2011 Dec 29. PMID 22209049
- [Background] Hou JM, Greystoke A, Lancashire L, Cummings J, Ward T, Board R, Amir E, Hughes S, Krebs M, Hughes A, Ranson M, Lorigan P, Dive C, Blackhall FH. Evaluation of circulating tumor cells and serological cell death biomarkers in small cell lung cancer patients undergoing chemotherapy. Am J Pathol. 2009 Aug;175(2):808-16. doi: 10.2353/ajpath.2009.090078. Epub 2009 Jul 23. PMID 19628770
- [Background] Hofman V, Long E, Ilie M, Bonnetaud C, Vignaud JM, Flejou JF, Lantuejoul S, Piaton E, Mourad N, Butori C, Selva E, Marquette CH, Poudenx M, Sibon S, Kelhef S, Venissac N, Jais JP, Mouroux J, Molina TJ, Vielh P, Hofman P. Morphological analysis of circulating tumour cells in patients undergoing surgery for non-small cell lung carcinoma using the isolation by size of epithelial tumour cell (ISET) method. Cytopathology. 2012 Feb;23(1):30-8. doi: 10.1111/j.1365-2303.2010.00835.x. Epub 2011 Jan 6. PMID 21210876
- [Background] Nieva J, Wendel M, Luttgen MS, Marrinucci D, Bazhenova L, Kolatkar A, Santala R, Whittenberger B, Burke J, Torrey M, Bethel K, Kuhn P. High-definition imaging of circulating tumor cells and associated cellular events in non-small cell lung cancer patients: a longitudinal analysis. Phys Biol. 2012 Feb;9(1):016004. doi: 10.1088/1478-3975/9/1/016004. Epub 2012 Feb 3. PMID 22306961
- [Background] Hofman V, Bonnetaud C, Ilie MI, Vielh P, Vignaud JM, Flejou JF, Lantuejoul S, Piaton E, Mourad N, Butori C, Selva E, Poudenx M, Sibon S, Kelhef S, Venissac N, Jais JP, Mouroux J, Molina TJ, Hofman P. Preoperative circulating tumor cell detection using the isolation by size of epithelial tumor cell method for patients with lung cancer is a new prognostic biomarker. Clin Cancer Res. 2011 Feb 15;17(4):827-35. doi: 10.1158/1078-0432.CCR-10-0445. Epub 2010 Nov 23. PMID 21098695
- [Background] Sawabata N, Okumura M, Utsumi T, Inoue M, Shiono H, Minami M, Nishida T, Sawa Y. Circulating tumor cells in peripheral blood caused by surgical manipulation of non-small-cell lung cancer: pilot study using an immunocytology method. Gen Thorac Cardiovasc Surg. 2007 May;55(5):189-92. doi: 10.1007/s11748-007-0101-2. PMID 17554991
- [Background] Sheu CC, Yu YP, Tsai JR, Chang MY, Lin SR, Hwang JJ, Chong IW. Development of a membrane array-based multimarker assay for detection of circulating cancer cells in patients with non-small cell lung cancer. Int J Cancer. 2006 Sep 15;119(6):1419-26. doi: 10.1002/ijc.21999. PMID 16642481
- [Background] Khoury S, Tran N. Circulating microRNAs: potential biomarkers for common malignancies. Biomark Med. 2015;9(2):131-51. doi: 10.2217/bmm.14.102. PMID 25689901
- [Background] Hofman V, Ilie MI, Long E, Selva E, Bonnetaud C, Molina T, Venissac N, Mouroux J, Vielh P, Hofman P. Detection of circulating tumor cells as a prognostic factor in patients undergoing radical surgery for non-small-cell lung carcinoma: comparison of the efficacy of the CellSearch Assay and the isolation by size of epithelial tumor cell method. Int J Cancer. 2011 Oct 1;129(7):1651-60. doi: 10.1002/ijc.25819. Epub 2011 Mar 11. PMID 21128227
- [Background] Went PT, Lugli A, Meier S, Bundi M, Mirlacher M, Sauter G, Dirnhofer S. Frequent EpCam protein expression in human carcinomas. Hum Pathol. 2004 Jan;35(1):122-8. doi: 10.1016/j.humpath.2003.08.026. PMID 14745734
- [Derived] Fu JY, Wen CT, Wu CF, Hsieh JC, Chang PC, Hsieh MJ, Liu YH, Lin YJ, Chang SC, Wu CY. Integrating Pathologic Stage and Perioperative Circulating Tumor Cell Variations: Early Relapse Prediction Model for Resectable Non-Small Cell Lung Cancer. JCO Precis Oncol. 2025 Apr;9:e2400709. doi: 10.1200/PO-24-00709. Epub 2025 Apr 28. PMID 40294350